CLINICAL TRIAL: NCT00903812
Title: A Retrospective and Prospective Observational Study Reviewing Supportive Care Management of NHL Patients Treated With CHOP-14 or 21 Chemotherapy(With or Without Rituximab) (CHOP = Cyclophosphamide, Hydroxyrubicin (Adriamycin), Oncovin (Vincristine), Prednisone Chemotherapy )
Brief Title: IMPACT Non Hodgkins Lymphoma (NHL) Study
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20060297
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2015-09

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: None Retained — This is an observational study. No bio-specimens are being collected.
  Time perspective - this study enrolls both retrospective and prospective subjects

GROUPS / COHORTS (1):
- A: No intervention - observational study
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention as observational study

SUMMARY:
This is multi-center, international observational study of subjects receiving CHOP-14 or CHOP-21 (with or without Rituximab) for the treatment of NHL. Approximately 100-150 sites will contribute information on subjects treated at their institution.

DETAILED DESCRIPTION:
This is a multi-center, international observational study of subjects receiving CHOP-14 or CHOP-21 (with or without Rituximab) for the treatment of NHL. Approximately 100-150 sites will contribute information on subjects treated at their institution.

To avoid geographical bias, sites will be selected to represent the spread of subjects in each country. Each site will be initially limited to 5 retrospective subjects and 10 prospective subjects (15 subjects per site) but sites may be asked to contribute further subjects to approximately 10 retrospective subjects and 20 prospective subjects.

Retrospective subjects may include any subject that has completed all cycles of chemotherapy treatment prior to date of site initiation. Prospective subjects which may be considered for the study are any subject planned for CHOP-14 or CHOP-21 (with or without Rituximab) treatment after the site initiation visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects greater than or equal to 18 years old
* Subjects diagnosed with any histological type of NHL (including both chemotherapy naïve and pre-treated subjects)
* Subjects planned to receive a minimum of 3 cycles of CHOP-14 or CHOP-21 with or without Rituximab (for subjects enrolled retrospectively, eligibility should be assessed on the profile at time of planning treatment, where treatment initiates on or after 01 Jan 2005, with specific focus on planned chemotherapy and not outcome or number of delivered cycles)
* Before any study-specific procedure, the appropriate written informed consent must be obtained for countries where this is required

Exclusion Criteria:

* Subjects receiving CHOEP ((CHOP = Cytoxan, Hydroxyrubicin (Adriamycin), Oncovin (Vincristine),Etoposide, Prednisone Chemotherapy )or CNOP (Cytoxan, Novantrone, Oncovin (Vincristine),Etoposide, Prednisone) chemotherapy are not eligible for inclusion in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects greater than or equal to 18 years old. Subjects diagnosed with any histological type of NHL (including both chemotherapy naïve and pre-treated subjects). Subjects planned to receive a minimum of 3 cycles of CHOP-14 or CHOP-21 with or without Rituximab (for subjects enrolled retrospectively, eligibility should be assessed on the profile at time of planning treatment, where treatment initiates on or after 01 Jan 2005, with specific focus on planned chemotherapy and not outcome or number of delivered cycles) . Before any study-specific procedure, the appropriate written informed consent must be obtained for countries where this is required
Sampling Method: Probability Sample
Enrollment: 1837 (Actual)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who had an investigator assessed risk of FN ≥20% and received primary prophylaxis G-CSF | At the end of observational period (when all subjects completed planned chemotherapy or stopped treatment)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Haioun C, Salar A, Pettengell R, Johnsen HE, Duehrsen U, Rossi FG, Verhoef G, Schwenkglenks M, Jaeger U, Hamilton L, Pujol B, Lugtenburg PJ. Anemia and erythropoiesis-stimulating agent administration in patients with non-Hodgkin lymphoma treated with cyclophosphamide, doxorubicin, vincristine, and prednisolone +/- rituximab chemotherapy: results from an observational study. Leuk Lymphoma. 2011 May;52(5):796-803. doi: 10.3109/10428194.2011.557166. Epub 2011 Feb 21. PMID 21338278
- [Background] Lugtenburg P, Silvestre AS, Rossi FG, Noens L, Krall W, Bendall K, Szabo Z, Jaeger U. Impact of age group on febrile neutropenia risk assessment and management in patients with diffuse large B-cell lymphoma treated with R-CHOP regimens. Clin Lymphoma Myeloma Leuk. 2012 Oct;12(5):297-305. doi: 10.1016/j.clml.2012.06.004. PMID 23040435
- [Background] Pettengell R, Johnsen HE, Lugtenburg PJ, Silvestre AS, Duhrsen U, Rossi FG, Schwenkglenks M, Bendall K, Szabo Z, Jaeger U. Impact of febrile neutropenia on R-CHOP chemotherapy delivery and hospitalizations among patients with diffuse large B-cell lymphoma. Support Care Cancer. 2012 Mar;20(3):647-52. doi: 10.1007/s00520-011-1306-6. Epub 2011 Nov 20. PMID 22101611
- [Background] Weycker D, Danel A, Marciniak A, Bendall K, Lipsitz M, Pettengell R. Economic costs of chemotherapy-induced febrile neutropenia among patients with non-Hodgkin's lymphoma in European and Australian clinical practice. BMC Cancer. 2012 Aug 22;12:362. doi: 10.1186/1471-2407-12-362. PMID 22913768
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com